CLINICAL TRIAL: NCT05949632
Title: A Phase 1/2 Study of INCB099280 in Combination With Axitinib in Adults With Advanced Solid Tumors
Brief Title: A Study of INCB099280 in Combination With Axitinib in Adults With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This was a strategic business decision. There were no safety concerns contributing to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB99280-201; 2023-510281-27-00 (Registry Identifier: EU CT Number); 2022-003663-13 (EudraCT Number)
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
Keywords: gynecologic tract cancer; ovarian cancer; primary peritoneum cancer; fallopian tube cancer; uterine cancer; cervical cancer; vulvar cancer; vaginal cancer; clear cell histology; mucinous adenocarcinoma; carcinosarcoma; serous adenocarcinoma; neuroendocrine histology; small cell histology; small-molecule pdl1 inhibitor; tyrosine kinase inhibitor; combination therapy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Adenocarcinoma, Mucinous; Carcinosarcoma; Cystadenocarcinoma, Serous | interventions — Axitinib

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts. In the Part 1 dose-escalation, participants will be enrolled in up to 6 dose levels of INCB099280 administered in combination with axitinib. In the Part 2 dose expansion, participants will be enrolled into 1 of 2 disease-specific cohorts at the dose(s) identified in Part 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: Dose Escalation (Experimental): Up to 6 doses of INCB099280 administered twice daily (BID) in combination with axitinib BID will be evaluated to identify dose(s) for further evaluation in the dose expansion phase of the study.
  Interventions: Drug: INCB099280; Drug: axitinib
- Part 2: Dose Expansion (Experimental): On completion of Part 1, participants will be enrolled in 1 of 2 disease-specific cohorts: Cohort 1: Adults with clear-cell gynecological cancers with at least 50% clear-cell histology whose disease progressed on or following at least 1 prior line of systemic chemotherapy and are not candidates for curative surgery or (chemo)radiation. Cohort 2: Adults with rare histological subtype epithelial cancers of the gynecological tract whose disease progressed on or following at least 1 prior line of systemic chemotherapy and are not candidates for curative surgery or (chemo)radiation. One or two doses may be selected from Part 1 for each cohort in the Part 2 Expansion.
  Interventions: Drug: INCB099280; Drug: axitinib

INTERVENTIONS:
Drug: INCB099280 — Administered as specified in the treatment arm description
Drug: axitinib — Administered as specified in the treatment arm description

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of INCB099280 in combination with axitinib and to assess the antitumor activity of INCB099280 in combination with axitinib. This study will only be open in the UK and EU.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumors (protocol-defined select solid tumors) with measurable lesions per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) that are considered non-amenable to surgery or other curative treatments or procedures.
* Must have disease progression on or after treatment with at least one prior systemic chemotherapy.
* Eastern Cooperative Oncology Group performance status score of 0 or 1.
* Life expectancy > 12 weeks.
* Willingness to avoid pregnancy.

Exclusion Criteria:

* Known additional malignancy that is progressing or requires active treatment.
* Central nervous system (CNS) metastases requiring treatment and/or leptomeningeal disease.
* Toxicity from prior therapy that has not recovered to protocol-defined limits.
* Prior receipt of an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent; treatment with an immune modulator (eg, CTLA-4, GITR, LAG3, TIM3, OX40, ICOS, IL-2, 4-1BB, CAR-T cell).
* Prior therapy with antiangiogenic small-molecule TKIs targeting the VEGF pathway
* Participation in another interventional clinical study while receiving INCB099280.
* Impaired cardiac function or clinically significant cardiac disease.
* History or evidence of interstitial lung disease including noninfectious pneumonitis.
* Presence of gastrointestinal conditions that may affect drug absorption.
* Any autoimmune disease requiring systemic treatment in the past 5 years.
* Diagnosis of primary immunodeficiency or receiving chronic systemic steroid therapy at a daily dose exceeding 10 mg of prednisone or equivalent.
* Active infection requiring systemic therapy.
* History of organ transplantation, including stem cell transplantation.
* Receipt of systemic antibiotics within 28 days of first dose of study treatment.
* Probiotic usage is prohibited during screening and throughout the study treatment period.
* Received a live vaccine within 28 days of the planned start of study drug.
* Laboratory values outside the Protocol-defined ranges.
* Inadequate organ function.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants with Dose Limiting Toxicities (DLTs) | Up to 21 days
  Dose-limiting toxicity will be defined as the occurrence of any of the toxicities as per protocol.
Part 1: Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years and 90 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Part 1: Number of participants with TEAEs leading to dose modification | Up to 2 years
  Number of participants with TEAEs leading to a dose modification (treatment interruption, dose reduction, and permanent discontinuation of either study drug).
Part 2: Objective response rate (ORR) | Up to 2 years
  Defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR), as determined by investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Part 2: Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years and 90 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Part 2: Number of participants with TEAEs leading to dose modification | Up to 2 years
  Number of participants with TEAEs leading to a dose modification (treatment interruption, dose reduction, and permanent discontinuation of either study drug).
Part 1: Objective response rate (ORR) | Up to 2 years
  Defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR), as determined by investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Disease Control Rate (DCR) | Up to 2 years
  Defined as the best overall response of CR, PR, or stable disease (SD) of at least 11 weeks from the start of treatment by investigator assessment per RECIST v1.1.
Duration of Response (DOR) | Up to 2 years
  Defined as the time from the first CR or PR until disease progression by investigator assessment per RECIST v1.1 or death from any cause, whichever occurs earlier.
INCB099280 and axitinib plasma concentrations. | Up to 2 years
  PK parameters will be calculated from the blood plasma concentrations of INCB099280 and axitinib using standard noncompartmental (model independent) PK methods.

CONTACTS AND LOCATIONS:
Overall Officials: Philomena Colucci, Study Director — Incyte Corporation
Locations (6):
- United Kingdom (6):
  - Addenbrookes Hospital, Cambridge
  - Beatson West of Scotland Cancer Centrewester, Glasgow
  - St Bartholomew'S Hospital, London
  - Guys Hospital, London
  - The Royal Marsden, London
  - The Royal Marsden Nhs Foundation Trust - Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency